CLINICAL TRIAL: NCT05091853
Title: Laparscopic Inguinal Hernia Repair - Does the Choice of Self-fixated Mesh Matter?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anna-Maria Thölix, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUS/3413/2020
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Inguinal Hernia; Surgery
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-adhesive mesh (Active Comparator)
  Interventions: Device: Adhesix mesh
- Self-gripping mesh (Active Comparator)
  Interventions: Device: Adhesix mesh

INTERVENTIONS:
Device: Adhesix mesh — 2 meshes are used; the self-gripping Progrip mesh and the self-adhesive Adhesix mesh
  Other Names: Progrip mesh

SUMMARY:
Self-fixed mesh and postoperative pain after laparoscopic inguinal hernia surgery, a randomized clinical trial

DETAILED DESCRIPTION:
Pain after inguinal hernia surgery is a major problem for the patient and results in lower quality of life. In this randomized clinical trial we examine if the choice of self-fixed mesh affects post-operative inguinal pain in laparoscopic hernia surgery. 164 patients are randomized and followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* patients with a clinical inguinal hernia, who are operated with laparoscopic surgery in day case surgery

Exclusion Criteria:

* scrotal or incarcerated hernia
* previous laparotomy
* ASA >3
* BMI <18 or >35
* Liver cirrhosis
* No hernia in clinical examination

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-05-09 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Pain during the first post-operative week | 1 year
  The degree of pain (VAS score) and the use of pain medication during the first postoperative week

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki ja uudenmaan sairaalhoitopiiri, Espoo, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tholix AM, Kossi J, Gronroos-Korhonen M, Harju J. Laparoscopic inguinal hernia repair with self-fixated meshes: a randomized controlled trial. Surg Endosc. 2025 Apr;39(4):2425-2435. doi: 10.1007/s00464-025-11616-5. Epub 2025 Feb 20. PMID 39979619